CLINICAL TRIAL: NCT01272128
Title: A Multicenter, Prospective Non-interventional Study to Evaluate the Quality of Life in Belgian Patients With CIS or RRMS in Whom Interferon Beta-1a IM Treatment Has Been Initiated
Brief Title: Avonex-evaluation of Quality of Life and Convenience in Belgian Participants - The AVAIL Study
Acronym: AVAIL
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: BE-AVO-01
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Interferon beta-1a — Interferon beta-1a will not be provided as a part of this study. Participants will receive Interferon beta-1a as prescribed by their treating physician prior to enrollment.
  Other Names: BG9418; Avonex Pen; Avonex

SUMMARY:
The primary objective is to assess the quality of life of intramuscular (IM) Interferon Beta-1a in participants with relapsing remitting multiple sclerosis (RRMS) or Clinically Isolated Syndrome (CIS) in a clinical practice setting.

ELIGIBILITY:
Key Inclusion Criteria:

* Decision to treat with Interferon Beta-1a (IFN beta-1a) must precede enrollment, independently of the study and in compliance with the marketing authorization
* Study enrollment must occur prior to 4th weekly administration of IFN beta-1a
* Able to understand and complete a self-administered questionnaire
* No contra-indications for IFN beta-1a

Key Exclusion Criteria:

* Subjects with history of hypersensitivity to natural or recombinant IFN beta or to any component
* Subjects with primary or secondary progressive MS
* Subjects with current severe depression and/or suicidal ideation
* Pregnant women
* Subjects participating in another clinical trial
* Subjects who do not want to participate in the study

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Relapsing Remitting Multiple Sclerosis (RRMS) or Clinically Isolated Syndrome (CIS) who meet the criteria for prescription of Interferon Beta-1a IM at up to 20 Belgian institutions may participate into this study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in EuroQol 5D (EQ-5D) Visual Analog Scale (VAS) at 12 months | Baseline and Month 12
  Quality of life will be assessed on a visual analog scale from 0 = worst imaginable health status to 100 = best imaginable health status.

SECONDARY OUTCOMES:
Change from Baseline in EQ-5D VAS at 6, 18 and 24 months | Baseline and Months 6, 18 and 24
  Quality of life will be assessed on a visual analog scale from 0 = worst imaginable health status to 100 = best imaginable health status.
Change from Baseline in the Multiple Sclerosis Impact Scale-29 (MSIS-29) score | Baseline and Months 6, 12, 18 and 24
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a patient-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a patient's perspective; it measures 20 physical items and 9 psychological items. The scores are generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.
Change from Baseline in EQ-5D Summary Score | Baseline and Months 6, 12, 18 and 24
  The EQ-5D is a self-administered questionnaire consisting of 5 questions pertaining to specific health states (i.e., mobility, self-care, pain/discomfort, usual activities and anxiety/depression), with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem). A summary index with a maximum score of 1 is derived from these five dimensions where a score of 1 indicates the best health state.
Convenience | Baseline and Months 6, 12, 18 and 24
  Convenience will be assessed by a self-administered convenience questionnaire that asks participants about their treatment satisfaction over the past 2 weeks.
Correlation between VAS and MSIS29 | Baseline and Months 6, 12, 18 and 24
  The correlation between the EQ-5D visual analog scale and Multiple Sclerosis Impact Scale 29 scores will be assessed using the Spearman correlation coefficient.
Correlation between VAS and Convenience questionnaire | Baseline and Months 6, 12, 18 and 24
  The correlation between the EQ-5D visual analog scale and convenience questionnaire results will be assessed using the Spearman correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (16):
- Belgium (16):
  - Research Site, Bonheiden, Antwerp
  - Research Site, Middelheim, Antwerp
  - Research Site, Ottignies, Brabant Wallon
  - Research Site, Woluwe, Brussels Capital
  - Research Site, Aalst, East Flanders
  - Research Site, Saint Niklaas, East Flanders
  - Research Site, Tielt, East Flanders
  - Research Site, Baudour, Hainaut
  - Research Site, Charleroi, Hainaut
  - Research Site, La Louvière, Hainaut
  - Research Site, Tournai, Hainaut
  - Research Site, Hasselt, Limburg
  - Research Site, Liège, Liège
  - Research Site, Verviers, Liège
  - Research Site, Libramont, Luxembourg
  - Research Site, Sijsele, West Flanders